CLINICAL TRIAL: NCT05558657
Title: Effect of Home-based Acupressure on Constipation in People with Spinal Cord Injury: a Study Protocol for a Randomized Controlled Trial with a Mixed-method Approach
Brief Title: Effect of Acupressure on Constipation in Community-dwelling Spinal Cord Injury Patients: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0035107
Record Dates: First submitted 2022-09-06; First posted 2022-09-28 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries; Traditional Chinese Medicine
Keywords: Spinal cord injury; Acupressure; Community-dwelling; Traditional Chinese Medicine
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: We aim to have two study group, including the intervention group that receive acupressure combined with nursing interventions, and the control group that receive acupressure on sham acupoints combined with nursing interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive home-based acupressure and nursing education.
  Interventions: Other: Home-based, acupressure combined with nursing education
- Control group: Home-based sham group , acupressure combined with nursing interventions (Active Comparator): The control group will receive home-based, manual light touch of the abdomen combined with nursing education.
  Interventions: Other: Home-based, manual light touch of the abdomen combined with nursing education

INTERVENTIONS:
Other: Home-based, acupressure combined with nursing education — The intervention group will focus on 11 acupoints on the abdomen (RN12, RN4, ST25), back (BL20, BL21, BL22, BL23, BL24, BL25), and limbs (LI4, ST36). The participants or their caregivers can perform acupressure 30 minutes after meals and twice a day. Participants can choose between two sets of acupressure: (1) Acupressure of the abdominal and back acupoints in a seated position, or (2) Acupressure of the abdominal and limb acupoints in a supine position. Each session lasts approximately 15 minutes.
  Besides, the intervention group will also receive nursing education on the basis of receiving acupressure intervention including (1) dietary guidance: help patients to formulate a reasonable diet plan, (2) cultivate regular defecation habits, (3) understand appropriate defecation environments and postures, and (4) Moderate exercise to increase gastrointestinal motility.
  Arms: Intervention group
Other: Home-based, manual light touch of the abdomen combined with nursing education — Control group or their caregivers will apply the manual light touch to the abdomen in any direction or body position at home. In keeping consistent with the intervention group, abdomen touching will also be administered twice daily for approximately 15 minutes each for 10 days. Participants will also receive nursing education.
  Arms: Control group: Home-based sham group , acupressure combined with nursing interventions

SUMMARY:
Spinal cord injury is a multi-sensory, motor and autonomic dysfunction, caused by various types of acute and chronic central nervous system injuries. And it will affect patient's ability to live normally and return to society. Due to lack of physical activity and psychological and environmental factors, the feces remain in the intestine for too long, and there will be excessive water absorption and lead to dryness and difficulty in excretion and it will be constipation. Chinese medicine, acupuncture and acupressure are the treatments of constipation in Traditional Chinese Medicine. Acupressure is a non- invasive intervention which is easy to learn and apply. We have carried out a number of studies on spinal cord injury rehabilitation support and acupressure to solve chronic problems such as constipation and anxiety. And this study aims to investigate the effects of acupressure combined with nursing intervention on constipation and quality of life in community-dwelling spinal cord injury patients.

DETAILED DESCRIPTION:
This study will use an open-label, double-group, randomized controlled trial to compare the effect of the intervention group with the control group. Study participants will be recruited from the "Hong Kong Direction Association for the Handicapped, a non-governmental organization dedicated to serving severely disabled Hong Kong people such as SCI. The sociodemographic data, disease status and outcome indicators of the study subjects were measured before the intervention, after the intervention and one month after the intervention. Research assistants (RA1) were trained to evaluate data and data, blinded to group assignments.

We will have the focus group interviews (semi-structured) with participants after the the intervention (post-intervention). The interviews will be conducted online to further understand the benefits and limitations of the research intervention.

ELIGIBILITY:
Inclusion Criteria:

1. being Hong Kong residents between the ages of 18 or older,
2. having an SCI diagnosis for over 6 months and living in the community,
3. demonstrating the willingness and ability to learn and engage in acupressure (or having a caregiver to assist if self-operating is not feasible),
4. experiencing difficulties with defecation or having concerns related to defecation.

Exclusion Criteria:

1. currently undergoing other TCM treatments or receiving interventions related to defecation or bowel functions,
2. being unable to attend the training sessions due to personal reasons,
3. having a history of gastrointestinal organic disease,
4. having severe metabolic diseases, cardiovascular, cerebrovascular, or mental illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The severity of constipation at baseline | The severity of constipation will be assessed at baseline assessment.
  Constipation Assessment Scale (CAS) will be used to measure the severity of constipation of the Spinal cord injury participants, 0 indicated no problem, 1 indicated some problem, 2 indicated severe problem. High scores will indicated the more severe condition of constipation.
The severity of constipation at post-intervention | The severity of constipation will be assessed after 10 days intervention.
  Constipation Assessment Scale (CAS) will be used to measure the severity of constipation of the Spinal cord injury participants, 0 indicated no problem, 1 indicated some problem, 2 indicated severe problem. High scores will indicated the more severe condition of constipation.
The severity of constipation at one month follow-up | The severity of constipation will be assessed after one month follow-up.
  Constipation Assessment Scale (CAS) will be used to measure the severity of constipation of the Spinal cord injury participants, 0 indicated no problem, 1 indicated some problem, 2 indicated severe problem. High scores will indicated the more severe condition of constipation.

SECONDARY OUTCOMES:
Quality of life at baseline | Quality of life will be assessed at baseline assessment.
  The Patient Assessment of Constipation Quality of Life Questionnaire will be used to measure the quality of life of Spinal cord injury participants. The scale investigates the quality of life of people in the past two weeks, using a 5-point Likert scale, assigning 0-4 points for various discomforts from "not at all" to "extremely". Each domain score and total score are the average scores of the domain items and all items, respectively. Higher scores indicate poorer quality of life.
Quality of life at post-intervention | Quality of life will be assessed after 10 days intervention.
  The Patient Assessment of Constipation Quality of Life Questionnaire will be used to measure the quality of life of Spinal cord injury participants. The scale investigates the quality of life of people in the past two weeks, using a 5-point Likert scale, assigning 0-4 points for various discomforts from "not at all" to "extremely". Each domain score and total score are the average scores of the domain items and all items, respectively. Higher scores indicate poorer quality of life.
Quality of life at one month follow-up | Quality of life will be assessed after one month follow-up.
  The Patient Assessment of Constipation Quality of Life Questionnaire will be used to measure the quality of life of Spinal cord injury participants. The scale investigates the quality of life of people in the past two weeks, using a 5-point Likert scale, assigning 0-4 points for various discomforts from "not at all" to "extremely". Each domain score and total score are the average scores of the domain items and all items, respectively. Higher scores indicate poorer quality of life.
Psychosocial well-being at baseline | Psychosocial well-being will be assessed at baseline assessment.
  The Depression Anxiety Stress Scale (DASS) will be used to measure participants' psychosocial well-being. The scale investigates the negative emotional experience or the corresponding physiological response in the last week.
Psychosocial well-being at post-intervention | Psychosocial well-being will be assessed after 10 days intervention.
  The Depression Anxiety Stress Scale (DASS) will be used to measure participants' psychosocial well-being. The scale investigates the negative emotional experience or the corresponding physiological response in the last week.
Psychosocial well-being at one month follow-up | Psychosocial well-being will be assessed after one month follow-up
  The Depression Anxiety Stress Scale (DASS) will be used to measure participants' psychosocial well-being. The scale investigates the negative emotional experience or the corresponding physiological response in the last week.
Bowel habit at baseline | Bowel habit will be assessed at baseline assessment.
  Bowel habits will be assessed during each visit by recording the frequency of laxative and glycerine enema use, as well as the frequency and duration of defecation in the past week.
Bowel habit at post-intervention | Bowel habit will be assessed after 10 days intervention.
  Bowel habits will be assessed during each visit by recording the frequency of laxative and glycerine enema use, as well as the frequency and duration of defecation in the past week.
Bowel habit at one month follow-up | Bowel habit will be assessed after one month follow-up.
  Bowel habits will be assessed during each visit by recording the frequency of laxative and glycerine enema use, as well as the frequency and duration of defecation in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Dr, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic Unviersity, Hong Kong, Hong Kong

REFERENCES:
- [Background] March, I.C.f.C.o.S.C.I.P.J.I., Global summary of spinal cord injury, incidence and economic impact. 2004.
- [Background] Qiu J. China Spinal Cord Injury Network: changes from within. Lancet Neurol. 2009 Jul;8(7):606-7. doi: 10.1016/S1474-4422(09)70162-0. No abstract available. PMID 19539234
- [Background] Zhao JR, Chen W, Zhao N, Zhang H. Q, Zhu. B. Research Progress on Mechanism of Traditional Chinese Medicine in Treatment of Spinal Cord Injury, Chinese Archives of Traditional Chinese Medicine. (2020); 8:1-14.
- [Background] Zhong C, Li YM. Overview of Chinese Medicine and Experimental Profiles on Spinal Cord Injury, Journal of Hunan University of Chinese Medicine. 2015; 35(10): 66-69.
- [Background] Sun Y, Zhan D, Tan MS, Discuss treating the Spinal Cord injury from the dredge of the Governor Vessel Chinese Journal of Traditional Medical Traumatology & Orthopedics. 2018; (2): 64-66.
- [Background] Sun Y. Study on the correlation between surgical treatment of atlantoaxial dislocation and nourishing qi and yang, Beijing University of Chinese Medicine. 2019.
- [Background] Xu W, Hao M. Clinical study on abdominal Eight Diagrams Manipulation Maneuver combined with nursing intervention in the treatment of constipation in patients with spinal cord injury, China Health Industry. 2013; 10(26): 190-191.
- [Background] Wong WK, Chien WT, Lee WM. Self-administered acupressure for treating adult psychiatric patients with constipation: a randomized controlled trial. Chin Med. 2015 Nov 3;10:32. doi: 10.1186/s13020-015-0064-7. eCollection 2015. PMID 26535053
- [Background] Liao CH, Xie ZL. Experience of traditional Chinese medicine nursing intervention on preventing constipation in bedridden patients with spinal cord injury experience, Chinese Community Doctors. 2012; 14(23): 299-300.
- [Background] Su SY, Qian R, Wei SH. Clinical observation of acupoint sticking in the treatment of constipation due to spleen deficiency and qi stagnation, Nei Mongol Journal of Traditional Chinese Medicine. 2018; 37(6): 96-97.
- [Background] Bengtsson M, Ohlsson B. Psychological well-being and symptoms in women with chronic constipation treated with sodium picosulphate. Gastroenterol Nurs. 2005 Jan-Feb;28(1):3-12. doi: 10.1097/00001610-200501000-00002. PMID 15738724
- [Background] De Giorgio R, Ruggeri E, Stanghellini V, Eusebi LH, Bazzoli F, Chiarioni G. Chronic constipation in the elderly: a primer for the gastroenterologist. BMC Gastroenterol. 2015 Oct 14;15:130. doi: 10.1186/s12876-015-0366-3. PMID 26467668
- [Background] Li HM, Gao JH. Clinical study of raw potato juice combined with abdominal Bagua massage in the treatment of spinal cord injury and constipation, Nei Mongol Journal of Traditional Chinese Medicine. 2014; 33(13): 37-38.
- [Background] Zhang D, Xia ZW. Rome III criteria for functional constipation, Chinese Journal of Medicine. 2008; 43(12): 63-64.
- [Background] Chang HC et al., Study on the effect of acupressure on constipation in nursing home residents, Journal of Yuanpei University. 2010; (17): 53-64.
- [Background] Chen YF. Effectiveness of the applying of acupressure and abdominal massage to improve constipation in stroke patients. 2017;1-146.
- [Background] Wang XD, Cai JP, Zhang YL. Effects of Xiao Zhang San on Umbilical Area Combined with the Acupoints Acupressure on Constipation, Nursing Journal of Chinese People's Liberation Army. 2013; 30(16).
- [Background] Chao ML, Chen LJ. Effects of Acupressure at Relieving Constipation in Persistent Vegetative State: A Randomized Controlled Trial, Journal of Integrated Chinese and Western Medicine. 2010; 12(2):11-20.
- [Background] Wang HP, et al., The effectiveness of Acupressure on Stroke Patents with Constipation, Chang Gung Nursing. 2006;17(4): 418-427.
- [Background] Xin LF, Pan YL. Effect of acupoint massage on preventing constipation in patients with cerebral hemorrhage, Chinese Journal of Modern Nursing. 2012; 18(22): 2699-2700.
- [Background] Chen XL, Wang YP. 50 cases of Acupoint massage of constipation in patients with senile dementia, Zhejiang Journal of Traditional Chinese Medicine. 2009; 44(2): 138-138.
- [Background] Lin SF, et al., Effectiveness of Acupressure on Elderly Patients with Constipation, Journal of Nursing and Healthcare Research. 2011; 7(3):175-187.
- [Background] Liao WF, Zhang H. Brief discussion on Tianshu Point, World Health Digest Medical Monthly. 2007; (4): p.139.
- [Background] Qin HB, Nan WZ, Yang M. General situation of clinical application of Zhongwan point, Hunan Journal of Traditional Chinese Medicine. 2018; 34(9): 214-216.
- [Background] Cheung DST, Tiwari A, Yeung WF, Yu DSF, So MKP, Chau PH, Wang XM, Lum TYS, Yuk Fung HYK, Ng BYM, Zhang ZJ, Lao L. Self-Administered Acupressure for Caregivers of Older Family Members: A Randomized Controlled Trial. J Am Geriatr Soc. 2020 Jun;68(6):1193-1201. doi: 10.1111/jgs.16357. Epub 2020 Feb 25. PMID 32096884
- [Background] Yeung WF, Ho FY, Chung KF, Zhang ZJ, Yu BY, Suen LK, Chan LY, Chen HY, Ho LM, Lao LX. Self-administered acupressure for insomnia disorder: a pilot randomized controlled trial. J Sleep Res. 2018 Apr;27(2):220-231. doi: 10.1111/jsr.12597. Epub 2017 Sep 8. PMID 28884877
- [Background] Chen YT, Chang YM, Bai CH. The Effectiveness of Acupressure at Relieving Constipation in Neurological Patients, Evidence Based Nursing. 2006; 2(4):301-310.
- [Background] Zhou RW, Traditional Chinese Medicine diagnosis of the Functional Constipation, Beijing Journal of Traditional Chinese Medicine. 2009; 28(2):115-116.
- [Background] Chen Z, et al., Clinical Study on Acupuncture at Jiaji Point for Spinal Cord Injury Constipation, Journal of Liaoning University of Traditional Chinese Medicine. 2014; 16(1): 189-190.
- [Background] McMillan SC, Williams FA. Validity and reliability of the Constipation Assessment Scale. Cancer Nurs. 1989 Jun;12(3):183-8. doi: 10.1097/00002820-198906000-00012. PMID 2743302
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Li Y, Bressington D, Chien WT. Pilot evaluation of a coping-oriented supportive program for people with spinal cord injury during inpatient rehabilitation. Disabil Rehabil. 2019 Jan;41(2):182-190. doi: 10.1080/09638288.2017.1386238. Epub 2017 Oct 10. PMID 28994618
- [Background] Li Y, Chien WT, Bressington D. Effects of a coping-oriented supportive programme for people with spinal cord injury during inpatient rehabilitation: a quasi-experimental study. Spinal Cord. 2020 Jan;58(1):58-69. doi: 10.1038/s41393-019-0320-2. Epub 2019 Jun 28. PMID 31253849
- [Background] Kwan RYC, Leung MCP, Lai CKY. A Randomized Controlled Trial Examining the Effect of Acupressure on Agitation and Salivary Cortisol in Nursing Home Residents with Dementia. Dement Geriatr Cogn Disord. 2017;44(1-2):92-104. doi: 10.1159/000478739. Epub 2017 Jul 29. PMID 28768251
- [Background] Chung KF, Yeung WF, Yu BY, Leung FC, Zhang SP, Zhang ZJ, Ng RM, Yiu GC. Acupuncture with or without combined auricular acupuncture for insomnia: a randomised, waitlist-controlled trial. Acupunct Med. 2018 Feb;36(1):2-13. doi: 10.1136/acupmed-2017-011371. Epub 2017 Dec 11. PMID 29229613
- [Derived] Li MQ, Li Y, Lam W, Yeung WF, Ho YS, Li JY, Sun TC, Yuen S, Hu YL, Yorke J. Home-based acupressure for managing constipation and subjective well-being in spinal cord injury survivors: A randomized controlled trial. J Integr Med. 2025 Nov;23(6):660-669. doi: 10.1016/j.joim.2025.08.001. Epub 2025 Aug 7. PMID 40846520